CLINICAL TRIAL: NCT03773640
Title: The Application of Radio Frequency Waves in Supportive Treatment of Temporomandibular Joint Dysfunction
Brief Title: The Application of Radio Frequency Waves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Malgorzata Pihut, Associate Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1072.6120.116.2018
Record Dates: First submitted 2018-12-09; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: temporomandibular joint dysfunction,; supportive treatment,; occlusal splint,; radiofreqency,; physiotherapy
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: The study group I (20 patients) and control group II (20 patients) consisted of patients, aged 19 to 45 years, of both sexes, who reported to the Consulting Room of Temporomandibular Joint Dysfunction at The Institute of Dentistry in Krakow to undertake prosthetic treatment of pain form of temporomandibular disorders, with the dominant muscle component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): Study group (I) consist of patients who were treated with the occlusal splints and radio frequency currents. In the case of application of radiation to the muscle area, the energy was 20 J and 15 J to the area of the masticatory muscles, the frequency was 3 MHz, bipolar technique, the duration of the procedure was 10 minutes, the coupling substance was a gel for ultrasound examinations.
  Interventions: Device: Radio frequency currents
- The control group (Active Comparator): The control group ( II) consisted of 20 patients treated with occlusion splints and sonophoresis procedures. For the area of mastication muscles 0.9 W/cm² treatments were applied, the duty factor was 80%, the treatment time was 10 minutes, and the medical substance was 25%Voltaren gel.
  Interventions: Drug: Sonophoresis

INTERVENTIONS:
Device: Radio frequency currents — Study group (I) consist of patients who were treated with the occlusal splints and radio frequency currents. In the case of application of radiation to the muscle area, the energy was 20 J and 15 J to the area of the masticatory muscles, the frequency was 3 MHz, bipolar technique, the duration of the procedure was 10 minutes, the coupling substance was a gel for ultrasound examinations.
  Arms: The study group
Drug: Sonophoresis — The control group ( II) consisted of 20 patients treated with occlusion splints and sonophoresis procedures. For the area of mastication muscles 0.9 W/cm² treatments were applied, the duty factor was 80%, the treatment time was 10 minutes, and the medical substance was 25%Voltaren gel.
  Arms: The control group

SUMMARY:
The aim of the study was to evaluate the influence of radio waves on the functioning of masseter muscles in the course of painful functional disorders of the organ, and thus the usefulness of these procedures in the treatment supporting temporomandibular joint dysfunction.

Material and method The study group I (20 patients) and control group II (20 patients) consisted of patients, aged 19 to 45 years, of both sexes, who reported to the Consulting Room of Temporomandibular Joint Dysfunction in Institute of Dentistry in Krakow to undertake prosthetic treatment of pain form of temporomandibular disorders with the dominant muscle component.

Study group (I) consist of patients who were treated with the occlusal splints and radio frequency currents. In the case of application of radiation to the muscle area, the energy was 20 J and 15 J to the area of the masticatory muscles, the frequency was 3 MHz, bipolar technique, the duration of the procedure was 10 minutes, the coupling substance was a gel for ultrasound examinations.

The control group ( II) consisted of 20 patients treated with occlusion splints and sonophoresis procedures. For the area of mastication muscles 0.9 W/cm² treatments were applied, the duty factor was 80%, the treatment time was 10 minutes, and the medical substance was 25%Voltaren gel.

DETAILED DESCRIPTION:
In recent years, the number of patients applying for prosthetic treatment due to painful forms of temporomandibular joint dysfunction has been increasing. Temporomandibular joints disorders (TMJD )include dysfunction of the masticatory muscles of the stomatognathic system, temporomandibular joints and the surrounding structures. There are often associated with abnormal conditions of occlusion.

The aim of the study was to evaluate the influence of radio waves on the functioning of masseter muscles in the course of painful functional disorders of the organ, and thus the usefulness of these procedures in the treatment supporting temporomandibular joint dysfunction.

Material and method The study group I (20 patients) and control group II (20 patients) consisted of patients, aged 19 to 45 years, of both sexes, who reported to the Consulting Room of Temporomandibular Joint Dysfunction in Institute of Dentistry in Krakow to undertake prosthetic treatment of pain form of temporomandibular disorders with the dominant muscle component.

Study group (I) consist of patients who were treated with the occlusal splints and radio frequency currents. In the case of application of radiation to the muscle area, the energy was 20 J and 15 J to the area of the masticatory muscles, the frequency was 3 MHz, bipolar technique, the duration of the procedure was 10 minutes, the coupling substance was a gel for ultrasound examinations.

The control group ( II) consisted of 20 patients treated with occlusion splints and sonophoresis procedures. For the area of mastication muscles 0.9 W/cm² treatments were applied, the duty factor was 80%, the treatment time was 10 minutes, and the medical substance was 25%Voltaren gel.

ELIGIBILITY:
Inclusion Criteria:

* pain form of temporomandibular joints dysfunction,
* the required age range,
* good general state of health,

Exclusion Criteria:

* the will (consent) of the patient,
* the presence of a general diseases,
* the presence of traumas,
* the presence of local inflammations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Assessment of intensity of pain (VAS - scale) | 10 weeks
  Assessment of intensity of pain of mastication muscles with the use of combined VAS and WNRS scales in own description.

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Department of Prosthetic Dentistry, Krakow, Lesser Poland Voivodeship, Poland